CLINICAL TRIAL: NCT00926861
Title: Posterior Macular Adhesion: A Potential Risk Factor for Non-exudative AMD to Develop Exudative AMD
Brief Title: Posterior Macular Adhesion: A Potential Risk Factor for Non-exudative Age Related Macular Degeneration (AMD) to Develop Exudative AMD
Acronym: PAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Ilse Krebs,MD, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Other Study IDs: 09-052-0409
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Dry Age-related Macular Degeneration; Detachment of the Posterior Hyaloid
Keywords: age-related macular degeneration; detachment of the posterior hyaloid; AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dry AMD: male or female persons aged over 50 years with dry age-related macular degeneration
  Interventions: Device: ultrasound; Device: OCT

INTERVENTIONS:
Device: ultrasound — A-scan and B-scan ultrasound at baseline and month 6,12,24
Device: OCT — Volume scans of spectralis OCT at baseline and month 6,12,24

SUMMARY:
Choroidal neovascularisation in age related macular degeneration is one of the major causes of legal blindness in the western world existing in two major occurences, the dry and the wet form.The etiology of age related macular degeneration is yet unknown. Genetic factors, oxidative stress, Ischaemia, and aging of the retinal pigment epithelium are discussed as etiologic factors. The risk of rapid vision loss is much higher in wet AMD, a dry form may transform to a wet form. From a prior study the investigators know that the posterior hyaloid is significantly more frequent attached in wet AMD. This study is conducted to examine whether the attached posterior hyaloid is a risk factor to develop wet AMD in dry AMD cases.

ELIGIBILITY:
Inclusion Criteria:

* Dry MD
* Age over 50 years

Exclusion Criteria:

* Macular pathologies other than age related macular degeneration (like diabetic maculopathy, macular pucker, macular hole)
* Prior vitrectomy or buckle surgery
* Uveitis posterior, multifocal chorioiditis
* Pathologic myopia
* Diabetic retinopathy
* Visualization of the macula not possible (dens cataract, vitreous haemorrhage)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female persons aged over 50 years with dry AMD
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Number of eyes with non-exudative AMD with attached and detached posterior vitreous cortex developing exudative AMD | 24 months

SECONDARY OUTCOMES:
Distance acuity | 24 months
Age | 24 months
Smoking | 24 months
Obesity | 24 months
Lesion classification (AREDS) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, Prof MD, Study Chair — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria